CLINICAL TRIAL: NCT06160973
Title: Food as Medicine for Families
Acronym: FAME-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Heart Association (Other); Community Servings (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 23-2420; 24RPGFIM1198190 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diet, Healthy; Loneliness
Keywords: Food Insecurity; Medically Tailored Meals; Nutrition Security

STUDY DESIGN:
Intervention Model Description: 2x2 Factorial Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Feed the household; Dedicated driver (Active Comparator): Medically tailored meals will be provided for the enrolled individual, with additional meals provided as needed for others living the same household; Medically tailored meals will be delivered each week by a driver who is an employee of Community Servings
  Interventions: Other: Feed the Household; Other: Dedicated Driver
- Feed the individual; Dedicated driver (Active Comparator): Medically tailored meals will be provided for the enrolled individual; Medically tailored meals will be delivered each week by a driver who is an employee of Community Servings
  Interventions: Other: Dedicated Driver; Other: Feed the Individual
- Feed the individual; Commercial shipper (Active Comparator): Medically tailored meals will be provided for the enrolled individual; Meals will be delivered by a commercial shipping organization
  Interventions: Other: Feed the Individual; Other: Commercial Shipper
- Feed the household; Commercial shipper (Active Comparator): Medically tailored meals will be provided for the enrolled individual, with additional meals provided as needed for others living the same household; Meals will be delivered by a commercial shipping organization
  Interventions: Other: Feed the Household; Other: Commercial Shipper

INTERVENTIONS:
Other: Feed the Household — Medically tailored meals will be provided for the enrolled individual, with additional meals provided as needed for others living the same household
  Arms: Feed the household; Commercial shipper; Feed the household; Dedicated driver
Other: Dedicated Driver — Medically tailored meals will be delivered each week by a driver who is an employee of Community Servings
  Arms: Feed the household; Dedicated driver; Feed the individual; Dedicated driver
Other: Feed the Individual — Medically tailored meals will be provided for the enrolled individual
  Arms: Feed the individual; Commercial shipper; Feed the individual; Dedicated driver
Other: Commercial Shipper — Meals will be delivered by a commercial shipping organization
  Arms: Feed the household; Commercial shipper; Feed the individual; Commercial shipper

SUMMARY:
The goal of this study is to determine the appropriate target of medically tailored meals (a particular individual vs. the entire household) and means of delivery (a dedicated delivery driver vs. a commercial shipper), to inform subsequent medically tailored meal trials.

DETAILED DESCRIPTION:
Medically tailored meals are thought to improve health by providing healthy foods, reducing food insecurity, and improving diet quality. However, there are two key open questions regarding implementation of medically tailored meals. One regards the 'target' of the intervention, and the other regards the mechanism of delivering the intervention. With regard to the target, there is an ongoing question about whether to provide meals for a specific individual only or for the entire household. Since food is shared in households, not feeding other household members could limit intervention effectiveness by 'underdosing' the intervention actually received by the target individual. Further, engaging in and sustaining healthy behavior change may be more difficult if others in the household are not involved, or if there is still not enough food to go around, resulting in ongoing household-level food insecurity despite the intervention. However, feeding the household is more expensive than feeding only a specific individual (although there are economies of scale). To date, medically tailored meal programs more commonly use a 'feed the individual' strategy, but some medically tailored meal organizations prefer a 'feed the household' strategy. Further, momentum is growing for a 'feed the household' strategy, perhaps best exemplified by Massachusetts' 1115 Waiver 'Flexible Services' re-authorization, the largest publicly funded medically tailored meal program in the country at the present time, which does include authorization to provide meals for the household in certain circumstances. Thus currently both strategies are in use by payers, though there is no evidence directly comparing them.

With regard to the delivery mechanism, medically tailored meals have historically been delivered by a member of the medically tailored meal organization. This personal connection is thought to have important benefits with regard to combating loneliness and social isolation, and features prominently as a mechanism of benefit in accounts from meal delivery organizations, prominently Meals on Wheels. However, shipping meals using commercial logistics firms (e.g., UPS) is likely less expensive and may allow reach into rural areas where a dedicated delivery driver may be cost prohibitive.

In this study, the investigators will conduct a 2x2 factorial randomized trial of 100 medically tailored meal participants in New England to help answer these questions. The first 'dimension' of the trial will test the impact of a 'feed the individual' vs. a 'feed the household' strategy for medically tailored meals. The second dimension will test the two methods of meal delivery (dedicated driver vs. commercial shipping). Key outcomes will be diet quality, loneliness, food security, and satisfaction with the program. The goal of this study is to determine the appropriate target of medically tailored meals and means of delivery, to inform subsequent medically tailored meal trials.

ELIGIBILITY:
Inclusion Criteria:

* No plans to move from the area for next 6 months
* Free living to the extent that participant has control over dietary intake
* Willing and able to provide written informed consent and participate in all study activities
* Able to complete study activities in English or Spanish

Exclusion Criteria:

* Lack of safe, stable residence and ability to store meals
* Lack of telephone
* Known psychosis or major psychiatric illness that prevents participation with study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Healthy Eating Index Total Score | 12 weeks
  Healthy Eating Index Score of diet quality, ranging from 0-100 with greater scores indicating greater diet quality. Derived from DietID assessments. This is the primary outcome for the 'feed the household' vs. 'feed the individual' aspect of the study.
De Jong Gierveld Total Loneliness Score | 12 weeks
  The 11-item De Jong Gierveld Total Loneliness instrument will be used. Scores range from 0 to 11 with greater scores indicating greater loneliness. This is the primary outcome for the 'dedicated driver' vs. 'commercial shipper' aspect of the study.

SECONDARY OUTCOMES:
Healthy Eating Index Subscores | 12 weeks
  13 subcomponents of the Healthy Eating Index Score of diet quality, ranging from 0-5, 0-10, or 0-20, with greater scores indicating greater diet quality. Derived from DietID assessments. These subscores are summed to yield the Healthy Eating Index Total Score
Dietary Screener Questionnaire (DSQ) Scores | 12 weeks
  Following current recommendations, the Dietary Screener Questionnaire results will be score to produce consumption estimates and other derived variables. In general, greater consumption of foods to be emphasized is associated with better health, and lower consumption of foods to be consumed in moderation is associated with better health.
  https://epi.grants.cancer.gov/nhanes/dietscreen/scoring/current/
Household Food Security Survey Module | 12 weeks
  The 18-item USDA Household Food Security Survey Module with 30-day lookback period will be administered. This will produce a raw score and categories of food insecurity, consistent with established scoring. https://www.ers.usda.gov/media/8271/hh2012.pdf
Health-Related Quality of Life | 12 weeks
  The EuroQol Five Dimension - Five Level (EQ-5D-5L) will be used to produce quality of life and health utility scores. Health utility scores range from 0 to 1, with 1 representing perfect health. https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/
Econ QOL Score | 12 weeks
  The Econ QOL Score will be used to capture economic quality of life. Resulting scores are on a T score metric (M=50, SD=10); higher scores indicate better economic quality of life
Depressive Symptoms | 12 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Depression 8a will be used to measure depressive symptoms. Greater scores indicate greater depressive symptoms.
De Jong Gierveld Emotional Loneliness Score | 12 weeks
  Scores range from 0 to 6 with greater scores indicating greater emotional loneliness
De Jong Gierveld Social Loneliness Score | 12 weeks
  Scores range from 0 to 5 with greater scores indicating greater social loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Berkowitz, MD MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC. These conditions are in addition to any funder requirements.
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC